CLINICAL TRIAL: NCT01210326
Title: The Comparison of Diagnostic Testicular Sperm Extraction(TESE) and Testicular Sperm Aspiration(TESA) in Non-obstructive Azoospermic Patients a Randomized Clinical Trial Study
Brief Title: The Comparison of Diagnostic TESE and TESA in Non-obstructive Azoospermic
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Hamid Gourabi,President of Royan institute, President of Royan Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Emb-009
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2008-08

CONDITIONS: Infertility
Keywords: TESE; TESA; non obstructive; azoospermi
MeSH Terms: conditions — Infertility | interventions — Sperm Retrieval

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aspiration (Experimental): 90 patients with non-obstructive azoospermi undergo testicular sperm aspiration
  Interventions: Procedure: testicular sperm aspiration
- extraction (Experimental): 90 patients with non-obstructive azoospermi undergo testicular sperm extraction
  Interventions: Procedure: extaction; Procedure: testicular sperm extraction

INTERVENTIONS:
Procedure: extaction — TESE (testicular sperm extraction), which is actually a surgical biopsy of the testis; or TESA (testicular sperm aspiration), which is performed by sticking a needle in the testis and aspirating fluid and tissue with negative pressure
  Other Names: Tecnique comparision
  Arms: extraction
Procedure: testicular sperm extraction — testicular sperm extraction
  Other Names: sperm extraction
  Arms: extraction
Procedure: testicular sperm aspiration — testicular sperm aspiration
  Other Names: sperm aspiration
  Arms: aspiration

SUMMARY:
Azoospermia , as the name suggests , refers to the condition in which there are no sperm in the semen. This diagnosis can come as a rude shock, because most men with a zero sperm count have normal libido; normal sexual function; and their semen looks completely normal too. The diagnosis can only be made by examining the semen under a microscope in the laboratory.Men with non-obstructive azoospermia have a normal passageway, but abnormal testicular function, and their testes do not produce sperm normally. Some of these men may have small testes on clinical examination. The testicular failure may be partial, which means that only a few areas of the testes produce sperm, but this sperm production is not enough for it to be ejaculated. Other men may have complete testicular failure, which means there is no sperm production at all in the entire testes. The only way to differentiate between complete and partial testicular failure is by doing multiple testicular micro-biopsies to sample different areas of the testes and send them for pathological examination. This technique is called TESA, or testicular sperm aspiration ( also known as TESE, or testicular sperm extraction) or mTESE ( micro-testicular sperm extraction).

DETAILED DESCRIPTION:
This study was performed on 180 men with non-obstructive azoospermia (NOA), referring to royan infertility center, according to inclusion and exclusion criteria. Testis selection (right and left) and techniques (TESE or TESA) were performed randomly in patients. For every patient based on random order, TESA or TESE was performed as the following procedures. The testis was aspirated at three separated sites (upper, middle and lower pole), using 20 ml syringe and 18-gauge needle or testicular biopsy (TESE) was taken from the same 3 sites.

ELIGIBILITY:
Inclusion Criteria:

* Non obstructive Azoospermia
* No Previous biopsy

Exclusion Criteria:

* Atrophic testis
* FSH levels more than 4 times normal range

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Sperm retrieval | 6 months
  comparision the success of sperm retrieval with TESE and TESA

SECONDARY OUTCOMES:
Side effects | 6 months
  Evaluate the side effects of the procedures like bleeding, inflammation, infection

CONTACTS AND LOCATIONS:
Overall Officials: hamid gourabi, PhD, Study Chair — President of Royan Institute; Jalil Hosseini, MD, Principal Investigator — urology investigator
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Royan Institute — http://www.royaninstitute.org